CLINICAL TRIAL: NCT03516721
Title: Chronotropic Incompetence During Exercise and Relations With Development of Cardiovascular Disease in Obese Adolescents
Brief Title: Chronotropic Incompetence During Exercise in Obese Adolescents: Clinical Implications and Pathophysiology
Acronym: CICO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hasselt University (Other)
Collaborators: Jessa Hospital (Other)
Responsible Party: Principal Investigator, Dominique Hansen, Principal Investigator, Hasselt University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: CICO-001
Record Dates: First submitted 2018-04-16; First posted 2018-05-04 (Actual); Last update posted 2020-02-11 (Actual); Status verified 2019-11

CONDITIONS: Obesity; Adolescent Obesity
MeSH Terms: conditions — Obesity; Pediatric Obesity | interventions — Clostridium perfringens epsilon-toxin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Obese adolescents (Other)
  Interventions: Other: the prevalence of chronotropic incompetence CI during maximal cardiopulmonary exercise testing, CPET
- Lean adolescents (Other)
  Interventions: Other: the prevalence of chronotropic incompetence CI during maximal cardiopulmonary exercise testing, CPET

INTERVENTIONS:
Other: the prevalence of chronotropic incompetence CI during maximal cardiopulmonary exercise testing, CPET

SUMMARY:
A reduction in peak heart rate (HR) and suppressed HR response during exercise is highly prevalent in obese populations. This phenomenon is also known as chronotropic incompetence (CI). In adult obese individuals, CI is independently related to elevated risk for major adverse cardiovascular events and premature death. Despite the established association between CI and prognosis in adult populations, the prognostic relevance of CI in adolescents with obesity has however deserved no attention, but is important. CI during exercise testing may indicate various, yet undetected anomalies, such as altered blood catecholamine and/or potassium concentrations during exercise, structural myocardial abnormalities or ventricular stiffness, impaired baroreflex sensitivity and cardiovascular autonomic dysfunction, atherosclerosis, or cardiac electrophysiological anomalies, which all have been detected in obese children and adolescents. However, whether CI during exercise testing may be a sensitive and specific indicator for these anomalies in obese adolescents has not been studied yet. In addition, the exact physiology behind obesity and development of heart disease remains to be studied in greater detail in obese adolescents. In this project, we examine the prevalence of CI (during maximal cardiopulmonary exercise testing, CPET) in 60 obese adolescents (aged 12-16 years) vs. 60 lean adolescents, and study the association between CI and changes in CPET parameters, lactate, catecholamine and potassium concentrations during CPET, biochemical variables, and cardiac electrophysiology (by ECG recording). In addition, the relation between CI and cardiac function (echocardiography) will be examined in a subgroup (29 lean and 29 obese) of these adolescents. In this regard, the diagnostic value of HR (responses) during maximal exercise testing will be clarified in obese adolescents, and the physiology behind the elevated risk for heart disease in obese adolescents can be explored.

ELIGIBILITY:
Inclusion Criteria:

* aged 12-16 years
* obese or lean (based on extended international (IOTF) body mass index cut-offs for thinness, overweight and obesity)
* Parental permission

Exclusion Criteria:

- Chronic cardiovascular, renal, pulmonary and orthopedic disease

Ages: 12 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 120 (Actual)
Dates: Start 2016-11-01 (Actual); Primary Completion 2017-05-01 (Actual); Study Completion 2019-08-31 (Actual)

PRIMARY OUTCOMES:
Heart rate (HR) | day 1
  Assessed using a 12-lead ECG device
Ventilatory function | day 1
  Determined during maximal cardiopulmonary exercise testing.

SECONDARY OUTCOMES:
height | day 1
weight | day 1
body composition | day 1
PAQ-A (Physical Activity Questionaire for Adolescents) | day1
  physical activity determined using the validated Dutch physical activity questionnaire for adolescents
Tanner scale | day 1
  Puberty stage (ranging from 1 to 5) will be assessed in all participants by the pediatric endocrinologist using Tanner staging criteria.
  Boys - development of external genitalia Girls - breast development Boys and girls - pubic hair
Plasma glucose | day 1
  blood analyses
iron | day 1
  blood analyses
aspartate aminotransferase | day 1
  blood analyses
alanine aminotransferase | day 1
  blood analyses
gamma-glutamyl transpeptidase | day 1
  blood analyses
alkaline phosphatase | day 1
  blood analyses
uric acid | day 1
  blood analyses
calcium | day 1
  blood analyses
blood total cholesterol | day 1
  blood analyses
high-density lipoprotein cholesterol | day 1
  blood analyses
low-density lipoprotein cholesterol | day 1
  blood analyses
proteins | day 1
  blood analyses
triglyceride concentrations | day 1
  blood analyses
c-reactive proteine | day 1
  blood analyses
thyroid-stimulating hormone | day 1
  blood analyses
free thyroxine | day 1
  blood analyses
cortisol and serum insulin | day 1
  blood analyses
serum leptin concentration | day 1
  blood analyses
blood haemoglobin | day 1
  blood analyses
haematocrit | day 1
  blood analyses
leukocytes | day 1
  blood analyses
Echocardiography | day 1
  Assessment left ventricular structure and systolic and diastolic function

CONTACTS AND LOCATIONS:
Overall Officials: Dominique Hansen, prof. dr., Principal Investigator — Hasselt University
Locations (1):
- Jessa Ziekenhuis, Hasselt, Belgium

IPD SHARING:
Plan to Share IPD: Undecided